CLINICAL TRIAL: NCT00575276
Title: Sex-Dependent Modulation of Clinical Outcomes Following Laparoscopic Cholecystectomy
Brief Title: Study of Pain Perception Between Males and Females Following Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kenneth Hargreaves, Chair Dept. of Endodontics, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC20070426
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Cholecystitis, Acute; Cholecystitis, Chronic
Keywords: Pain, Cholecystectomy, Cytokines, Sex Differences
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1 cm biopsies of the body and fundus of the excised gallbladder. Two 4ml blood samples collected for DNA analysis with future studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Females with acute cholecystitis
- 2: Females with Chronic Cholecystitis
- 3: Males with acute cholecystitis
- 4: Males with Chronic Cholecystitis

SUMMARY:
This study looks at the differences in inflammatory mediators in gallbladder tissue between males and females and the possibility that these differences contribute to a higher perception of post-operative pain in females following laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
A patient's gender is a strong and significant predictor for substantial differences in clinical outcomes such as postoperative pain, analgesic use, and surgical complications (gangrenous gallbladder, empyema of the gallbladder, gallbladder perforation, and conversion to open surgery) following laparoscopic cholecystectomy (Bingener et al., 2002; Bingener et al., 2003; Uchiyama et al., 2006). Although females present for laparoscopic cholecystectomy more frequently (76% of the cases); the prevalence of surgical complications during cholecystectomy is higher in men, most frequently because of inflammation or deterioration of the gallbladder (Bingener et al., 2002; Bingener et al., 2003; Stefanidis et al., 2006). Post-operatively, however, females report significantly greater pain scores and require larger amounts of analgesics (Uchiyama et al., 2006), suggesting that although surgeries are completed with fewer problems, females still report more post-operative pain. Sex-related differences in pain thresholds and tolerance to thermal, pressure, and electrical stimuli in experimental pain models indicate that pain differences are not solely due to psychosocial distinctions between the sexes (Riley et al., 1998).

There are multiple physiological differences between males and females; however, considerable evidence implicates estrogenic sex hormones as critical factors in sex-dependent differences in pain (see review by Fillingim and Ness, 2000). It is possible that estrogens alter inflammatory mediator profiles in the gallbladder, which subsequently increase sensitization of visceral neurons innervating the gallbladder, resulting in increased pain in females. The first portion of this study will extend the association of patient sex with clinical outcomes to determine whether circulating and/or local estrogen levels correlate with differences in peri-operative morbidity, including intra-operative complications, conversion to open cholecystectomy, postoperative pain, inadequate wound healing, intra-abdominal infection, disability and mortality.

Previous studies have demonstrated that the cytokines TNFalpha and IL-1beta alter the sensitivity of sensory neurons and increase nociception (Opree and Kress, 2000). To determine whether estrogen levels alter the profile of inflammatory mediators within the gallbladder and result in an increase in nociceptive thresholds in females, we will correlate circulating and/or local levels of estrogens with the amount of inflammatory mediators present within laparoscopically excised gallbladder biopsies. Patients who meet the inclusion criteria will be recruited from University Hospital in San Antonio. Inflammatory mediators, including the cytokines IL-1beta, TNFalpha, IL-8, IL-6, IL-10, and IL-12p70 will be assayed from interstitial fluid of biopsies from the fundus and infundibulum of the gallbladder. Biopsies will be classified according to clinical assessment prior to surgery to control for expected differences in inflammatory mediators in acute versus chronic cholecystitis.

The immediate effects of this research will be to clearly delineate whether estrogens are predictive of improved clinical outcomes following surgery and to determine whether these sex hormones correlate with altered production of inflammatory mediators in the gallbladder.

ELIGIBILITY:
Inclusion Criteria:

* Males or Non-pregnant females
* Between ages 18-90

Exclusion Criteria:

* Pregnant Females within six months of surgery
* Individuals below age 18 or above age 90
* Previous topical or systemic corticosteroid use within three months of surgery date
* sign and symptoms of neuropathy or self-reported history of diseases or treatments known to be associeated with neuropathy
* signs and symptoms of altered immune system or self-reported diseases or treatments known to be associated with altered immune function

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient General Surgery patients indicated for Laparoscopic Cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2006-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Hargreaves, DDS, PhD, Principal Investigator — University of Texas Health Science Center San Antonio; Juliana Bingener-Casey, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University Hospital System, San Antonio, Texas, United States